CLINICAL TRIAL: NCT03626532
Title: Mind-body Interventions for Healthy Aging
Acronym: HealthyAgers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Ruchika Prakash, Associate Professor - Clinical, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017H0223; R01AG054427 (NIH)
Record Dates: First submitted 2018-08-04; First posted 2018-08-13 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Aging
Keywords: Mindfulness-based stress reduction; Cognitive function; Emotion regulation; Lifestyle education; Attentional control; Mindfulness training; Aging; Older adults; Mind-wandering; Functional connectivity; Randomized controlled trial
MeSH Terms: conditions — Emotional Regulation | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single-blind. Any investigators administering assessments will be blind to participants' group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Stress Reduction (Experimental): Participants will meet once a week for 8 weeks (2.5 hours per session), plus a 4-hour retreat day, to engage in mindfulness meditation exercises. Didactic components will include oral presentations, informational videos, and group discussion. Additionally, daily homework assignments will require participants to engage in guided practices for 30 minutes a day for 5 days a week.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR)
- Lifestyle Education (Active Comparator): Participants will meet once a week for 2.5 hours for 8 weeks, plus a 4-hour retreat day, to engage in light stretching exercises and interactive discussions on health topics, such as physical activity, nutrition, sleep, stress, etc. Didactic components will include oral presentations, informational videos, and group discussion. Additionally, daily homework assignments will ask participants to engage in stretching, read or watch informational content, and answer reflection questions for 30 minutes a day for 5 days a week.
  Interventions: Behavioral: Lifestyle Education (LifeEd)

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MBSR) — The MBSR program is a mind-body approach developed by Kabat-Zinn to reduce pain and stress through mindfulness meditation. MBSR is a form of mental training characterized by the self-regulation of attention and focal orientation to present moment experiences. Mindfulness practice is thought to effectively promote emotional and cognitive control. Mindfulness includes directing awareness away from thoughts, emotions and sensations towards some specific "anchor" to the present, such as the breath. Participants will engage in various practices including breath awareness, body scans, mindful listening, etc.
  Other Names: MBSR
  Arms: Mindfulness-Based Stress Reduction
Behavioral: Lifestyle Education (LifeEd) — This group will engage in light stretching exercises at each session. They will also be provided with information drawn from the scientific literature on topics related to healthy aging, including physical activity, sedentary behavior, nutrition, hydration, stress, sleep, and cognitively stimulating activities. Group discussion will be incorporated throughout.
  Other Names: LifeEd
  Arms: Lifestyle Education

SUMMARY:
The goal of this study is to examine the impact of mind-body interventions in enhancing behavioral and neural correlates of attentional control in older adults. Participants will be randomized to either a 8-week mindfulness meditation group or a 8-week lifestyle education group. Additional booster sessions, spanning the course of a year, will be offered to participants in both groups. Participants will complete pre- and post-assessments of neurocognitive and emotional functioning, and will be assessed for maintained benefits 12-months post-intervention.

DETAILED DESCRIPTION:
Mind-body interventions are increasingly being examined for their potential to improve cognitive function, enhance emotion regulation, reduce stress and related inflammatory markers, and alter the neural circuitry supporting cognitive and emotional functioning. The primary goal of this study is to examine changes in attentional control resulting from engaging in mind-body interventions with additional booster sessions over the course of a year. Within this goal, the behavioral and neural mechanisms of change in attentional control will be investigated and the transfer of benefits to performance on measures of everyday cognition and emotion regulation will be assessed. Our main hypothesis is that eight weeks of mindfulness training will increase attentional control performance in the elderly, partially through mindfulness-induced reductions in mind-wandering and changes in the functional architecture of the brain. Up to 200 older adults (ages 65-85) will be enrolled for the study. Of these, 151 older adults meeting eligibility criteria will be randomized to either an eight-week MBSR (mindfulness based stress reduction) program or a lifestyle education group. Participants will attend weekly mindfulness training or lifestyle education sessions and will be asked to complete homework assignments administered via a mobile/web-based application designed by the laboratory. All participants will also be invited to participate in four booster sessions over the course of 12 months following the intervention with continued access to the mobile application content. Behavioral metrics of cognitive function and inflammatory markers will be collected before and after the eight-week intervention as well as at 6-months and 12-month follow-up assessments. Neural metrics of cognitive functioning will be collected before and after the eight-week intervention as well as at 12-month follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 65-85 years
* Capable of attending the assessment and the majority of intervention sessions
* Right-handed
* Fluent English speaker
* Corrected (near and far) visual acuity of 20/40 or better
* Normal color vision
* Adequate hearing for experimental purposes
* Absence of diagnosed terminal illness
* Absence of diagnosed neurological disorders
* No history of psychotic disorder or substance abuse disorder
* Absence of any psychiatric disorder that was 1) diagnosed by a psychologist or psychiatrist and 2) diagnosed within the past 2 years OR symptoms and/or treatment is ongoing
* Score less than 20 on the Center for Epidemiologic Studies Depression Scale (CES-D)
* Absence of medication use that significantly alters brain activity
* No history of diagnosed learning disability that would interfere with the completion of cognitive tasks
* No evidence of dementia: No scores below 2 standard deviations from the mean on neuropsychological battery AND adequate self-reported performance of instrumental activities of daily living
* To be included in the MRI portion of the study (not exclusionary for study participation): Absence of any non-MRI safe objects that cannot be removed, not pregnant and not attempting to become pregnant, and absence of self-reported claustrophobia
* Able to engage in light stretching exercises with or without assistive devices
* No regular practice of meditation or yoga (defined as once or more per week) AND no previous participation in a structured mindfulness class such as MBSR
* Access to the internet

Exclusion Criteria:

* Not between the ages of 65-85
* Any physical limitation or pragmatic limitation that prohibits attendance at assessment sessions and intervention sessions
* Left-handed or ambidextrous
* No fluency in English
* Corrected (near or far) visual acuity worse than 20/40
* All types of color blindness
* Self-reported hearing impairment that would affect their ability to hear the experimenter
* Diagnosis of terminal illness
* Presence of diagnosed neurological disorders
* History of psychotic disorder or substance abuse disorder diagnosed by a psychologist or psychiatrist
* History of psychotic disorder or substance abuse disorder diagnosed by a psychologist of psychiatrist
* Presence of any psychiatric disorder that was 1) diagnosed by a psychologist or psychiatrist and 2) diagnosed within the past 2 years OR symptoms/treatment is on going
* Score greater than or equal to 20 on the CES-D
* Medication use that significantly alters brain activity
* History of diagnosed learning disability that would interfere with completion of the cognitive tasks
* Evidence of dementia: one or more memory scores below 2 standard deviations from the mean AND one or more non-memory scores below 2 standard deviations from the mean on neuropsychological battery OR total score below 2 standard deviations from the mean on neuropsychological battery OR inadequate self-reported performance of instrumental activities of daily living
* Presence of non-MRI safe objects that cannot be removed, pregnant or attempting to become pregnant, or self-reported claustrophobia (exclusionary for MRI portion of the study only)
* Actual or perceived limitation that prohibits engaging in light stretching exercises with or without assistive devices
* Any regular practice of meditation or yoga (defined as once or more per week) OR previous participation in a structured mindfulness class such as MBSR
* No access to the internet

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 173 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Change in attentional control on tasks of sustained attention | Baseline, 2 months, 8 months, 14 months
  Participants will complete computerized measures of Continuous Performance Test and Go/No-Go Task to assess sustained attention. Detectability (d') measures will be calculated to assess the effects of mind-body interventions on attentional control. Data collected at 8-months and 14-month will be used to determine maintenance effects.

SECONDARY OUTCOMES:
Change in neural functioning during measures of attentional control | Baseline, 2 months, 14 months
  Participants will complete an functional magnetic resonance imaging (fMRI) assessment before and after the intervention. Functional connectivity changes will be examined during tasks of attentional control to determine neural correlates of mind-body interventions.
Change in mind-wandering on tasks of sustained attention | Baseline, 2 months, 8 months, 14 months
  To measure mind-wandering, participants will also be prompted with quasi-random probes asking them to categorize the thoughts they were having immediately preceding the probe.
Change in emotion regulation strategy sse | Baseline, 2 months, 8months, 14 months
  Participants will complete lab-based and ecological momentary assessment (EMA)-based emotion regulation strategy use tasks to determine change in ER strategy use following mind-body interventions.
Change in cognitive performance on the NIH Cognitive Toolbox Battery | Baseline, 2 months, 8 months, 14 months
  Participants will perform the NIH Cognitive Toolbox Battery comprised of seven different tasks aimed at measuring episodic memory, executive function, attention, working memory, language, and processing speed. Change on this measure will be assessed to determine the impact of the mind-body interventions on various domains of cognitive functioning.
Change in Measure of Daily Functioning | Baseline, 2 months, 8 months, 14 months
  Participants will complete the Driving Scenes subtest of the Neuropsychological Assessment Battery (NAB) as a measure of everyday cognition. This subtest measures attention and working memory to changing driving scenes.
Change in inflammatory biomarkers | Baseline, 2 months, 8 months, 14 months
  Data on inflammatory markers - C-reactive protein (CRP), interleukin 6 (IL-6), and interleukin 10 (IL-10) - will be collected to determine the impact of mind-body interventions on systemic markers of inflammation.
Change in self-report measures of stress | Baseline, 2 months, 8 months, 14 months
  Participants will be administered the Perceived Stress Scale (PSS) to measure changes in self-reported perceived stress following mind-body interventions. This measure has 10 items, each measured on a 5-point rating scale. One total score will be calculated by summing the individual item responses. Higher scores represent greater feelings of stress, unpredictability, and uncontrollability.
Change in self-report measures of emotion dysregulation | Baseline, 2 months, 8 months, 14 months
  Participants will be administered the Difficulties in Emotion Regulation Scale (DERS) to examine changes in degree of self-reported emotion dysregulation following mind-body interventions. This measure has 36 items, each measured on a 5-point rating scale. One total score will be calculated by summing the individual item responses. Higher scores represent greater perceived difficulties in emotion regulation capabilities.
Change in self-report measures of quality of life | Baseline, 2 months, 8 months, 14 months
  Participants will be administered the The World Health Organization Quality of Life abbreviated scale (WHOQOL-BREF) to examine changes in self-reported quality of life following mind-body interventions. This measure has 26 items, each measured on a 5-point rating scale. Four domains are measured by taking the average of representative items: psychological (six items), environmental (eight items), physical health (seven items), and social relationships (three items), as well as overall QoL (two items). Higher scores represent better perceived quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ruchika Prakash, Ph.D., Principal Investigator — The Ohio State Universty
Locations (1):
- Department of Psychology, The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prakash RS, Fountain-Zaragoza S, Fisher M, Gbadeyan O, Andridge R, Kiecolt-Glaser J, Manglani HR, Duraney EJ, Shankar A, McKenna MR, Teng J, Phansikar M, Canter R. Protocol for a randomized controlled trial of mindfulness-based stress reduction to improve attentional control in older adults (HealthyAgers trial). BMC Geriatr. 2022 Aug 13;22(1):666. doi: 10.1186/s12877-022-03334-7. PMID 35964000